CLINICAL TRIAL: NCT01578434
Title: Role of Calcium And Vitamin D In Nutritional Rickets And It's Management
Acronym: ROCAVINR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Varun, Principal Investigator, Senior Resident Physician, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rickets 1
Record Dates: First submitted 2012-04-12; First posted 2012-04-17 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Nutritional Rickets
Keywords: Nutritional Rickets; Calcium; Vitamin D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D; Calcium Carbonate; Calcium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Calcium Carbonate (Active Comparator): Calcium: 75 mg/kg calcium daily for 3 months
  Interventions: Drug: Calcium Carbonate
- Vitamin D (Active Comparator): Vitamin D: 6 lakh IU single im dose
  Interventions: Drug: Vitamin D
- Vitamin D and Calcium (Active Comparator): vitamin D and Calcium: combination of above two
  Interventions: Drug: Vitamin D and Calcium

INTERVENTIONS:
Drug: Vitamin D — Vitamin D: 6 lakh IU single im dose Calcium: 75 mg/kg calcium daily for 3 months vitamin D and Calcium: combination of above two
  Arms: Vitamin D
Drug: Calcium Carbonate — Calcium: 75 mg/kg calcium daily for 3 months
  Arms: Calcium Carbonate
Drug: Vitamin D and Calcium — Vitamin D: 6 lakh IU single im dose. along with Calcium: 75 mg/kg calcium daily for 3 months
  Arms: Vitamin D and Calcium

SUMMARY:
Rickets, a common nutritional disorder, is usually considered to be due to vitamin D deficiency. However, in the last few decades many studies have shown that in tropical countries, with abundance of sunshine, calcium deficiency may play a more important role in the causation of rickets. Studies from adults in India have also shown that calcium intake of our population is much below the recommended allowance. The calcium deficiency gets compounded by the high level of phytates in the conventional vegetarian diet consumed by the majority of the population. There are few studies on children in India / other Asian countries on assessment of dietary calcium intake.

However, recent studies from many nations of the world have also shown a wide spread prevalence of vitamin D deficiency in adolescent and adult population. A study done at our own hospital has shown a high prevalence of vitamin D deficiency in lactating mothers and their infants.

Since both Calcium and Vitamin D deficiency are likely to be present in children, it is not clear what plays a more important role in the etiology of rickets in India or other Asian countries.

The present study is therefore planned with the following objectives:

1. To study the dietary calcium intake, sun exposure and serum vitamin D levels in children with and without rickets.
2. To compare the role of Calcium Carbonate, Vitamin D and a combination of the two in the treatment of nutritional rickets.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6 months to 5 years with rickets

Exclusion Criteria:

* Non nutritional cause of rickets
* taken vitamin D or calcium supplements in last 6 months
* children presenting with convulsions

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2007-11; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Healing of rickets | 6 months
  Assessment of healing of rickets on biochemical and radiological assessment